CLINICAL TRIAL: NCT01026272
Title: Quantification of Novel Immune Markers in Human Serum of Patients With MS
Brief Title: Novel Immune Markers in Patients With Multiple Sclerosis
Acronym: NIMMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Michelle Sexton ND, University of Washington
Other Study IDs: 35083-B; A50879 (Other: University of Washington)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Sclerosis
Keywords: Endocannabinoid; Fish Oil; Multiple Sclerosis; Monocyte Migration
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy subjects: subjects with no sign of inflammatory disease, or diagnosis of MS
- Patients with MS

SUMMARY:
The investigators hypothesize that the endogenous cannabinoid signalling system has lost homeostasis in the disease multiple sclerosis (MS). To investigate a novel action of dietary fish oils, the investigators will administer a food frequency questionnaire to both healthy subjects and patients with MS. The investigators will first determine if there are differences between both populations of endogenous cannabinoids, and then determine whether dietary intake of fish oils alters these levels

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for MS patients:

1. Diagnosis of Multiple Sclerosis (relapsing, remitting) made by a clinical neurologist within the previous 5 years by either MRI (> 3 white matter lesions) or score of 3-5 on the Kurtzke Expanded Disability Status Scale.
2. Not currently in "relapse" or exacerbation.
3. Age > 21 and < 50.
4. Subjects must be able to attend study visits at screening, baseline and time points of 4, 12 and 24 weeks.
5. Diet, exercise, and supplementation must be kept constant throughout participation in the study.
6. Ability to read and speak English.

Inclusion criteria for healthy subjects:

1. Current.
2. Age > 21 and < 50.
3. Subjects must be able to attend study visits at screening, baseline and time points 4, 12 and 24 weeks.
4. Diet, exercise, and supplementation must be kept constant throughout participation in the study.
5. Ability to read and speak English.

Exclusion Criteria:

1. Supplementation with fish oils in the last six months.
2. Diagnosis of any bleeding disorder (hemophilia, vonWillebrands, menorrhagia, hypercoaguability, history of clots, thrombocytopenia). Any patient with one of these diagnoses and/or any patient on any of/combination of the following medications would not be eligible for participation: ANTICOAGULANT/ANTIPLATELET DRUGS: Some of these drugs include aspirin, clopidogrel (Plavix), dalteparin (Fragmin), dipyridamole (Persantine), enoxaparin (Lovenox), heparin, ticlopidine (Ticlid), warfarin (Coumadin).
3. Hormone Replacement Therapy or oral contraception pills or pregnancy.
4. Use of clinical Cannabis for MS symptom control or recreationally in the last 6 months.
5. Previous diagnosis of DSMV criteria.
6. Use of tobacco, either orally or inhaled.
7. BMI >27 or <19.
8. Diagnosis of Diabetes (fasting blood sugar over 125 mg/dl).
9. Performance athletes.
10. Medical history/diagnosis of autoimmune or other chronic inflammatory disease or serious immunologically-related health condition.
11. Lactose intolerance (in-ability to eat/drink milk products without problems).
12. Allergy to fish or seafood. Theoretically, some people who are allergic to seafood such as fish might also be allergic to fish oil supplements. There is no reliable information showing how likely people with seafood allergy are to have an allergic reaction to fish oils; however, until more is known advise patients allergic to seafood to avoid or use fish oil supplements cautiously.
13. High dose supplement/botanical therapy which may have an effect on bleeding times: Vitamin E (greater than 400 IU/qd); adn/or daily use of any/combination of the following botanical therapy: Angelica sinensis; Allium sativum; Zingiber officinale; Ginkgo biloba; and Salix alba.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Multiple Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Quantification of endogenous cannabinoids | one time blood draw

SECONDARY OUTCOMES:
Monocyte migration | one time blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Sexton, ND, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States